CLINICAL TRIAL: NCT00506649
Title: Comparison of no Protocol vs Protocolized Approach to Pain, Sedation and Delirium Management in the ICU
Brief Title: Improved ICU Outcomes With Protocolized Management of Analgesia, Sedation and Delirium
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Other Study IDs: 007
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Critical Care
Keywords: protocol; analgesia; sedation; delirium; coma
MeSH Terms: conditions — Agnosia; Delirium; Coma | interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: protocol — management protocols of non-pharmacological strategies and individualized titration of analgesics, sedatives, and anti-psychotics based on observed scores to manage sedation, analgesia and delirium.

SUMMARY:
To assess pain, agitation, and delirium experienced by critically ill patients daily and evaluate the impact of a protocol; to compare the incidence of coma and delirium, length of stay, mortality and costs of care between pre- and post-protocol groups.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to ICU

Exclusion Criteria:

* Repeat admission within the same hospitalisation; moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1214 (Actual)
Dates: Start 2003-08; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoanna Skrobik, MD FRCP(c), Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hopital Maisonneuve Rosemont, Montreal, Quebec, Canada